CLINICAL TRIAL: NCT01806207
Title: A Double-blind, Randomized, Multi-centre Study of the Efficacy and Safety of a Single Intra-articular Injection With Durolane Compared to Saline in Patients With Unilateral Knee Osteoarthritis
Brief Title: Durolane Compared to Saline in Patients With Unilateral Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35GA0301
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2013-03

CONDITIONS: Unilateral Knee Osteoarthritis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Durolane injection (Active Comparator): Intraarticular injection of 3 ml Durolane.
  Interventions: Device: Durolane injection
- Saline injection (Placebo Comparator): Intraarticular injection of physiological sodium chloride (0.9% NaCl) solution pH 7.
  Interventions: Other: Saline injection

INTERVENTIONS:
Device: Durolane injection
  Arms: Durolane injection
Other: Saline injection
  Arms: Saline injection

SUMMARY:
This was a study that compared Durolane injections to saline injections in the treatment of unilateral osteoarthritis of the knee. The patients were randomly assigned one of the two treatments unaware of which treatment they received. The study was conducted at 13 centers in Germany, the United Kingdom and Sweden. Patients were followed for six weeks after study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis according to ACR (American College of Radiology) criteria for the knee
* WOMAC pain score in the range 7 to 17
* Significant knee pain for the majority of days during the past 3 months
* Patient normally active, not bedridden or confined to a wheelchair and able to walk 50 meters without the help of a walker, crutches or a cane
* Patient has attempted but not responded adequately to non-pharmacological therapy(ies)
* Patient co-operative and able to communicate effectively with the investigators
* Signed informed consent obtained

Exclusion Criteria:

* Bilateral knee osteoarthritis
* Osteoarthritis or clinically significant pain from other part of the musculoskeletal system than the study knee
* Kellgren Lawrence radiographic score grade IV for the study knee
* Change in physical therapy/occupational therapy for the knee within the last 3 months
* Treatment with nonsteroidal antiinflammatory drugs (NSAIDs) (including topical agents for the study knee) during the last week (or 5 half-lives of the drug, whichever is longer) prior to baseline visit
* Treatment with non-NSAID topicals such as capsaicin for the knee within the last 3 days
* Intra-articular injection with corticosteroids in the study knee within the last 3 months
* Use of systemic steroids (excluding inhalation steroids) within the last 3 months
* Intra-articular injections with hyaluronic acid in the study knee within the last 9 months
* Treatment with glucosamine/chondroitin sulfate within the last 3 months
* Treatment with pain relievers except for paracetamol up to 4g/day
* Treatment with anticoagulant (except for acetylsalicylic acid max. 325 mg/day)
* Arthroscopy or any other surgical procedure in the study knee within the last 12 months
* Planned arthroscopy or any other surgical procedure during the study period
* Any medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion (e.g. severe progressive chronic disease, malignancy, bleeding disorder, fibromyalgia)
* Systemic active inflammatory condition or infection, such as Rheumatoid arthritis, inflammatory arthritis, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, gout/acute pseudogout or any other connective tissue disease
* Septic arthritis in the study knee within the last 3 months
* Active skin disease or infection in the area of the injection site
* Significant venous or lymphatic stasis present in the legs
* Pregnant or breast-feeding woman or woman of child-bearing potential not practicing adequate contraception
* Subjects that in the opinion of the investigator are unsuitable for inclusion (e.g. subjects not likely to avoid other therapies, subjects not likely to stay in the study during the whole study period, or subjects likely to be unreliable)
* Concurrent participation in any other clinical study or participation within the preceding 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2003-02; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Proportion of responders at 6 weeks. | At 6 weeks after treatment
  Proportion of responders was based on the improvement in WOMAC (Western Ontario and McMasters Universities Osteoarthritis Index) pain score.

SECONDARY OUTCOMES:
WOMAC pain score | 2 and 4 weeks after treatment
Safety of intraarticular injections of 3 ml Durolane | Through 6 weeks after treatment
  Safety was assessed by adverse event soliciting.
WOMAC stiffness score | 2, 4 and 6 weeks after treatment
WOMAC physical function score | 2, 4 and 6 weeks after treatment
Patient assessed global status | 2, 4 and 6 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Arden, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southhampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Arden NK, Akermark C, Andersson M, Todman MG, Altman RD. A randomized saline-controlled trial of NASHA hyaluronic acid for knee osteoarthritis. Curr Med Res Opin. 2014 Feb;30(2):279-86. doi: 10.1185/03007995.2013.855631. Epub 2013 Nov 5. PMID 24168077